CLINICAL TRIAL: NCT01525316
Title: Lactoferrin for Prevention of Sepsis in Infants
Acronym: NEOLACTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIDISI 57710; 1R01HD067694-01A1 (NIH)
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Late Onset Neonatal Sepsis
Keywords: Late Onset Neonatal Sepsis; Neonates; Lactoferrin; Infections; Prevention; Neurodevelopment
MeSH Terms: conditions — Neonatal Sepsis; Infections | interventions — Lactoferrin; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bovine Lactoferrin (Experimental): Lactoferrin is a freeze-dried protein purified directly from fresh bovine milk.
  Interventions: Dietary Supplement: Bovine Lactoferrin
- Maltodextrin (Placebo Comparator): Maltodextrin is an inert sugar.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Bovine Lactoferrin — Infants will receive oral bovine lactoferrin (200 mg/Kg/day divided in three dosis) for 8 weeks. Lactoferrin will be dissolved in human milk or infant formula or in a 5% glucose solution. Each dose will be dissolved in a small volume so the maximum lactoferrin concentration will be 25mg/mL.
  Other Names: Lactoferrin
  Arms: Bovine Lactoferrin
Dietary Supplement: Maltodextrin — Infants will receive oral maltodextrin (200mg/Kg/day in three divided dosis) for 8 weeks. Maltodextrin will be dissolved in human milk or infant formula or in a 5% glucose solution. Each dose will be dissolved in a small volume so the maximum maltodextrin concentration will be 25mg/mL.
  Arms: Maltodextrin

SUMMARY:
The investigators propose a clinical trial in premature infants to determine the effect of orally-administered bovine lactoferrin on occurrence of severe infections and to determine whether as a result of decreased infections, infants' growth and development improve after daily lactoferrin supplementation, due to its antimicrobial and anti-inflammatory properties. If successful, the use of lactoferrin as a protective protein could profoundly affect clinical care of neonates both in the developed and developing world.

DETAILED DESCRIPTION:
Neonatal mortality is an important global public health challenge. Approximately 4 million neonatal deaths per year occur in developing countries, accounting for 40% all of deaths in children under 5. Infection, birth asphyxia and consequences of premature birth/low birth weight are responsible for the majority of these deaths. Although advances in neonatal intensive care led to improved survival of premature infants, sepsis continues to be an important cause of morbidity and mortality worldwide.

Lactoferrin, an iron-binding protein with multiple physiological functions (anti-microbial, anti-inflammatory, and immunomodulatory), is one of the most important proteins present in mammalian milk. Our hypothesis is that lactoferrin given as a daily oral food supplement to preterm infants will improve their health by mimicking its protective role in milk. There is a vast literature showing in vitro and animal model benefits of lactoferrin. However, there are few clinical studies designed to translate this knowledge into patient care. A recent Italian study showed that lactoferrin given to low-birth weight infants reduces incidence of sepsis (17% vs. 6%) and death. Whether lactoferrin has an effect in higher risk populations and an impact on subsequent neurodevelopment and growth remains to be determined.

Specific aim 1: The investigators will test the hypothesis that bovine lactoferrin supplementation prevents serious infections in preterm infants. The investigators will conduct a randomized placebo-controlled double blind study in 414 premature infants < 2000 g in Neonatal Units in Lima, Peru to determine whether bovine lactoferrin prevents late-onset sepsis or sepsis-associated death.

This hypothesis is based on lactoferrin´s antimicrobial and immunomodulating activities. Lactoferrin protects against pathogens in multiple ways: it sequesters iron essential for bacterial growth; binds to lipopolysaccharide (LPS) on the cell surface of Gram negative bacteria, disrupting the bacterial cell membrane; it has anti-lipoteichoic acid (against Gram positive organisms) and anti-Candida cell wall activities. The investigators have found that lactoferrin not only inhibits growth; it impairs virulence of some of the major pathogens by decreasing their ability to adhere or to invade mammalian cells, and by binding to, or degrading, specific virulence proteins. Lactoferrin may protect infants from sepsis by blocking attachment and invasion of organisms in the gut.

Specific aim 2: The investigators will test the hypothesis that bovine lactoferrin supplementation promotes better neurodevelopment and growth outcomes in preterm infants assessed by the Mullen Scales of Early Learning, a standardized neurologic exam and growth measurements at 12, 18 and 24 months corrected age.

It is postulated that exposure of the preterm brain to inflammatory mediators during infectious episodes contribute to brain (white matter) injury and poor developmental outcome. It has been demonstrated that breast milk has a beneficial effect on neurodevelopment outcomes in preterm infants. The investigators hypothesize that lactoferrin is the major factor in milk responsible for this effect due to its antimicrobial and immunomodulatory properties: it reduces inflammation by decreasing production of tumor necrosis factor α and other pro-inflammatory molecules, and by regulating the immune response, protecting against severe inflammation related to infection and septic shock. In addition, the investigators hypothesize that lactoferrin will improve growth by decreasing the frequency of growth-impairing infections and by lactoferrin effect on intestinal cell proliferation, differentiation and maturation.

The use of lactoferrin as a broad-spectrum non-pathogen specific antimicrobial protective protein is an innovative approach. If successful this study will profoundly affect clinical care of neonates both in the developed and developing world.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with a birth weight between 500g and 2000g
* Neonates born in, or referred to the Neonatal Intermediate and Intensive Care Units of one of the participating hospitals in the first 72 hours of life.

Exclusion Criteria:

* Neonates with underlying gastrointestinal problems that prevent oral intake.
* Neonates with predisposing conditions that profoundly affect growth and development (chromosomal abnormalities, structural brain anomalies, severe congenital abnormalities).
* Neonates who have a family history of cow milk allergy.
* Neonates that, according to the investigator criteria, will not have the chance to complete the subsequent study visits (patients that before one month old would not be living in Lima).
* Neonates whose parents decline to participate.

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 414 (Actual)
Dates: Start 2012-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
First episode of late-onset sepsis or sepsis-associated death | 72hrs to 8 weeks of age
  The primary study outcome will be a composite outcome of the first episode of late-onset sepsis or sepsis-associated death.

SECONDARY OUTCOMES:
Neurodevelopment | 12 to 24 months of corrected age
  Neurodevelopment at 24 months of corrected age, assessed by the Mullen Scale for Early Learning.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa J Ochoa, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (3):
- Peru (3):
  - Hospital Nacional Alberto Sabogal Sologuren, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima

REFERENCES:
- [Background] Manzoni P, Rinaldi M, Cattani S, Pugni L, Romeo MG, Messner H, Stolfi I, Decembrino L, Laforgia N, Vagnarelli F, Memo L, Bordignon L, Saia OS, Maule M, Gallo E, Mostert M, Magnani C, Quercia M, Bollani L, Pedicino R, Renzullo L, Betta P, Mosca F, Ferrari F, Magaldi R, Stronati M, Farina D; Italian Task Force for the Study and Prevention of Neonatal Fungal Infections, Italian Society of Neonatology. Bovine lactoferrin supplementation for prevention of late-onset sepsis in very low-birth-weight neonates: a randomized trial. JAMA. 2009 Oct 7;302(13):1421-8. doi: 10.1001/jama.2009.1403. PMID 19809023
- [Background] Ochoa TJ, Zegarra J, Cam L, Llanos R, Pezo A, Cruz K, Zea-Vera A, Carcamo C, Campos M, Bellomo S; NEOLACTO Research Group. Randomized controlled trial of lactoferrin for prevention of sepsis in peruvian neonates less than 2500 g. Pediatr Infect Dis J. 2015 Jun;34(6):571-6. doi: 10.1097/INF.0000000000000593. PMID 25973934
- [Background] Akin IM, Atasay B, Dogu F, Okulu E, Arsan S, Karatas HD, Ikinciogullari A, Turmen T. Oral lactoferrin to prevent nosocomial sepsis and necrotizing enterocolitis of premature neonates and effect on T-regulatory cells. Am J Perinatol. 2014 Dec;31(12):1111-20. doi: 10.1055/s-0034-1371704. Epub 2014 May 16. PMID 24839144
- [Derived] Torres Roldan VD, Urtecho S M, Gupta J, Yonemitsu C, Carcamo CP, Bode L, Ochoa TJ. Human milk oligosaccharides and their association with late-onset neonatal sepsis in Peruvian very-low-birth-weight infants. Am J Clin Nutr. 2020 Jul 1;112(1):106-112. doi: 10.1093/ajcn/nqaa102. PMID 32401307
- [Derived] Ochoa TJ, Zegarra J, Bellomo S, Carcamo CP, Cam L, Castaneda A, Villavicencio A, Gonzales J, Rueda MS, Turin CG, Zea-Vera A, Guillen D, Campos M, Ewing-Cobbs L; NEOLACTO Research Group. Randomized Controlled Trial of Bovine Lactoferrin for Prevention of Sepsis and Neurodevelopment Impairment in Infants Weighing Less Than 2000 Grams. J Pediatr. 2020 Apr;219:118-125.e5. doi: 10.1016/j.jpeds.2019.12.038. Epub 2020 Feb 6. PMID 32037149
- [Derived] Medina-Alva P, Duque KR, Zea-Vera A, Bellomo S, Carcamo C, Guillen-Pinto D, Rivas M, Tori A, Zegarra J, Cam L, Castaneda A, Villavicencio A, Ochoa TJ. Combined predictors of neurodevelopment in very low birth weight preterm infants. Early Hum Dev. 2019 Mar;130:109-115. doi: 10.1016/j.earlhumdev.2019.01.019. Epub 2019 Feb 8. PMID 30743197
- [Derived] Rueda MS, Calderon-Anyosa R, Gonzales J, Turin CG, Zea-Vera A, Zegarra J, Bellomo S, Cam L, Castaneda A, Ochoa TJ; NEOLACTO Research Group. Antibiotic Overuse in Premature Low Birth Weight Infants in a Developing Country. Pediatr Infect Dis J. 2019 Mar;38(3):302-307. doi: 10.1097/INF.0000000000002055. PMID 29613975
- [Derived] Turin CG, Zea-Vera A, Rueda MS, Mercado E, Carcamo CP, Zegarra J, Bellomo S, Cam L, Castaneda A, Ochoa TJ; NEOLACTO Research Group. Lactoferrin concentration in breast milk of mothers of low-birth-weight newborns. J Perinatol. 2017 May;37(5):507-512. doi: 10.1038/jp.2016.265. Epub 2017 Jan 26. PMID 28125095